CLINICAL TRIAL: NCT03240328
Title: The Effect of CAR-T Cell Therapy on the Reconstitution of HIV-specific Immune Function
Brief Title: The Effect of Chimeric Antigen Receptor (CAR)-T Cell Therapy on the Reconstitution of HIV-specific Immune Function
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Guangzhou 8th People's Hospital (Other)
Collaborators: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Linghua LI, Vice Chief physician, Guangzhou 8th People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20170407V3
Record Dates: First submitted 2017-05-21; First posted 2017-08-07 (Actual); Last update posted 2022-09-14 (Actual); Status verified 2022-09

CONDITIONS: HIV/AIDS
Keywords: CAR-T HIV therapy; immunotherapy; function cure
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Immunotherapy, Adoptive

STUDY DESIGN:
Intervention Model Description: No control.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CAR-T therapy (Experimental): Transfusing CAR-T cells at least 1 million clone every time (once or twice) based on cART after attaining plasma HIV suppression (plasma HIV RNA <50 cp/ml) and CD4+ cell count more than 350 cells/ul over 1 year by cART without active HCV or HBV infection or opportunistic infections. If the candidates reach the criteria of discontinuing cART, they will stop cART and receive close observation. Once the plasma HIV viral load rebound to over 1000 cp/ml, they will restart cART immediately.
  Interventions: Biological: CAR-T cells

INTERVENTIONS:
Biological: CAR-T cells — HIV-1 specific chimeric antigen receptor cells

SUMMARY:
To study the safety and effectiveness of CAR-T Cell therapy on HIV patients whose plasma HIV has been successfully suppressed after cART, which is expected to enhance the res-constitution of HIV-specific immune function to assist the eradication of HIV reservoir.

DETAILED DESCRIPTION:
Despite the advent of combined antiretroviral therapy (cART), the persistence of viral reservoirs remains a major barrier to curing human immunodeficiency virus type 1 (HIV-1) infection. Recently, the shock and kill strategy, by which HIV-1 reservoirs could be eradicated following reactivation of latent HIV-1 by latency-reversing agents (LRAs), has been extensively practiced. It is important to reestablish virus-specific and reliable immune surveillance to eradicate the reactivated virus-harboring cells.the VC-CAR-T cells effectively induced the cytolysis of LRA-reactivated HIV-1-infected CD4 T lymphocytes isolated from infected individuals receiving successful cART. Our previous study demonstrated that the special features of genetically engineered CAR-T cells make them a particularly suitable candidate for therapeutic application in efforts to reach a functional HIV cure. In this clinical trial, we intend to study the safety and effectiveness of CAR-T Cell Therapy on HIV patients whose plasma HIV has been successfully suppressed after cART, by observing the adverse events, HIV-1 reservoir and the immune index.

ELIGIBILITY:
Inclusion Criteria:

1. HIV infection confirmed.
2. Receiving cART more than 12 months.
3. HIV viral-load < 50 copies/ml and CD4 cell count more than 350 cells/ul.
4. Without serious liver, heart, liver and kidney diseases.
5. The subjects know about the study and volunteer to attend the research and sign the informed consent.

Exclusion Criteria:

1. With active HBV or HCV infection, or serious opportunistic infections.
2. With serious chronic disease such like diabetes, the mental illness,et al
3. History of suffering from pancreatitis during cART.
4. Pregnant or breast-fed.
5. With poor adherence.
6. Unable to complete follow up.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-10-04 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-associated adverse events of CAR-T cell therapy | 6 Months
  To observe the adverse events of VC-CAR-T cell therapy on HIV-infected patients during the clinical trial

SECONDARY OUTCOMES:
HIV-1 reservoir | 6 Months
  To assay the HIV loads in the peripheral blood Mono-nuclear cells and plasma
HIV viral load rebound time | 6 months
  To assay the HIV viral load rebound period after discontinuing cART

OTHER OUTCOMES:
HIV-specific immunity | 6 Months
  To assay the remaining concentration of VC-CAR-T cells in patients, the number of HIV-specific CD4,CD8 and their activity after receiving CAR-T cell therapy

CONTACTS AND LOCATIONS:
Overall Officials: Cai Weiping, Bachelor, Principal Investigator — Guangzhou 8th People's Hospital
Locations (1):
- Guangzhou 8th People's Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Grupp SA, Kalos M, Barrett D, Aplenc R, Porter DL, Rheingold SR, Teachey DT, Chew A, Hauck B, Wright JF, Milone MC, Levine BL, June CH. Chimeric antigen receptor-modified T cells for acute lymphoid leukemia. N Engl J Med. 2013 Apr 18;368(16):1509-1518. doi: 10.1056/NEJMoa1215134. Epub 2013 Mar 25. PMID 23527958
- [Background] Kochenderfer JN, Dudley ME, Feldman SA, Wilson WH, Spaner DE, Maric I, Stetler-Stevenson M, Phan GQ, Hughes MS, Sherry RM, Yang JC, Kammula US, Devillier L, Carpenter R, Nathan DA, Morgan RA, Laurencot C, Rosenberg SA. B-cell depletion and remissions of malignancy along with cytokine-associated toxicity in a clinical trial of anti-CD19 chimeric-antigen-receptor-transduced T cells. Blood. 2012 Mar 22;119(12):2709-20. doi: 10.1182/blood-2011-10-384388. Epub 2011 Dec 8. PMID 22160384
- [Background] Lee DW, Kochenderfer JN, Stetler-Stevenson M, Cui YK, Delbrook C, Feldman SA, Fry TJ, Orentas R, Sabatino M, Shah NN, Steinberg SM, Stroncek D, Tschernia N, Yuan C, Zhang H, Zhang L, Rosenberg SA, Wayne AS, Mackall CL. T cells expressing CD19 chimeric antigen receptors for acute lymphoblastic leukaemia in children and young adults: a phase 1 dose-escalation trial. Lancet. 2015 Feb 7;385(9967):517-528. doi: 10.1016/S0140-6736(14)61403-3. Epub 2014 Oct 13. PMID 25319501
- [Background] Chimeric Antigen Receptor-Modified T Cells in Chronic Lymphoid Leukemia; Chimeric Antigen Receptor-Modified T Cells for Acute Lymphoid Leukemia; Chimeric Antigen Receptor T Cells for Sustained Remissions in Leukemia. N Engl J Med. 2016 Mar 10;374(10):998. doi: 10.1056/NEJMx160005. No abstract available. PMID 26962747
- [Background] Kochenderfer JN, Rosenberg SA. Chimeric antigen receptor-modified T cells in CLL. N Engl J Med. 2011 Nov 17;365(20):1937-8; author reply 1938. doi: 10.1056/NEJMc1111004. No abstract available. PMID 22087695
- [Background] Romeo C, Seed B. Cellular immunity to HIV activated by CD4 fused to T cell or Fc receptor polypeptides. Cell. 1991 Mar 8;64(5):1037-46. doi: 10.1016/0092-8674(91)90327-u. PMID 1900456
- [Background] Sahu GK, Sango K, Selliah N, Ma Q, Skowron G, Junghans RP. Anti-HIV designer T cells progressively eradicate a latently infected cell line by sequentially inducing HIV reactivation then killing the newly gp120-positive cells. Virology. 2013 Nov;446(1-2):268-75. doi: 10.1016/j.virol.2013.08.002. Epub 2013 Sep 6. PMID 24074590
- [Background] Ni Z, Knorr DA, Bendzick L, Allred J, Kaufman DS. Expression of chimeric receptor CD4zeta by natural killer cells derived from human pluripotent stem cells improves in vitro activity but does not enhance suppression of HIV infection in vivo. Stem Cells. 2014 Apr;32(4):1021-31. doi: 10.1002/stem.1611. PMID 24307574
- [Background] MacLean AG, Walker E, Sahu GK, Skowron G, Marx P, von Laer D, Junghans RP, Braun SE. A novel real-time CTL assay to measure designer T-cell function against HIV Env(+) cells. J Med Primatol. 2014 Oct;43(5):341-8. doi: 10.1111/jmp.12137. Epub 2014 Aug 20. PMID 25138734
- [Background] Zhen A, Kamata M, Rezek V, Rick J, Levin B, Kasparian S, Chen IS, Yang OO, Zack JA, Kitchen SG. HIV-specific Immunity Derived From Chimeric Antigen Receptor-engineered Stem Cells. Mol Ther. 2015 Aug;23(8):1358-1367. doi: 10.1038/mt.2015.102. Epub 2015 Jun 8. PMID 26050990
- [Background] Liu L, Patel B, Ghanem MH, Bundoc V, Zheng Z, Morgan RA, Rosenberg SA, Dey B, Berger EA. Novel CD4-Based Bispecific Chimeric Antigen Receptor Designed for Enhanced Anti-HIV Potency and Absence of HIV Entry Receptor Activity. J Virol. 2015 Jul;89(13):6685-94. doi: 10.1128/JVI.00474-15. Epub 2015 Apr 15. PMID 25878112
- [Background] Dotti G, Gottschalk S, Savoldo B, Brenner MK. Design and development of therapies using chimeric antigen receptor-expressing T cells. Immunol Rev. 2014 Jan;257(1):107-26. doi: 10.1111/imr.12131. PMID 24329793
- [Result] Liu B, Zou F, Lu L, Chen C, He D, Zhang X, Tang X, Liu C, Li L, Zhang H. Chimeric Antigen Receptor T Cells Guided by the Single-Chain Fv of a Broadly Neutralizing Antibody Specifically and Effectively Eradicate Virus Reactivated from Latency in CD4+ T Lymphocytes Isolated from HIV-1-Infected Individuals Receiving Suppressive Combined Antiretroviral Therapy. J Virol. 2016 Oct 14;90(21):9712-9724. doi: 10.1128/JVI.00852-16. Print 2016 Nov 1. PMID 27535056
- [Derived] Liu B, Zhang W, Xia B, Jing S, Du Y, Zou F, Li R, Lu L, Chen S, Li Y, Hu Q, Lin Y, Zhang Y, He Z, Zhang X, Chen X, Peng T, Tang X, Cai W, Pan T, Li L, Zhang H. Broadly neutralizing antibody-derived CAR T cells reduce viral reservoir in individuals infected with HIV-1. J Clin Invest. 2021 Oct 1;131(19):e150211. doi: 10.1172/JCI150211. PMID 34375315